CLINICAL TRIAL: NCT06780150
Title: SurfSubQ - A Prospective Longitudinal Multicenter Observational Study to Investigate Neurofilament Light Chain Levels and Patient Satisfaction After Subcutaneous Ocrelizumab Administration in Persons With Multiple Sclerosis
Brief Title: A Study to Investigate Effects of Ocrelizumab Treatment on Neurofilament Light Chain (NfL) Levels and Participant Satisfaction in Participants With Multiple Sclerosis (MS)
Acronym: SurfSubQ
Status: Recruiting | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML45551
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ocrelizumab: Participants who are receiving ocrelizumab, SC injection, for the first time as part of their routine MS therapy at physician's discretion in accordance with local clinical practice and/or labeling will be observed for treatment satisfaction with SC injection for up to 12 months.
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — Ocrelizumab will be administered as SC injection as per discretion of the treating physician in accordance with local clinical practice and local labeling.
  Other Names: RO4964913, Ocrevus

SUMMARY:
The main purpose of the study is to evaluate participant satisfaction after administration of ocrelizumab subcutaneous (SC) after 12 months using the therapy administration satisfaction questionnaire subcutaneous (TASQ-SC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS
* RMS and PPMS participants diagnosed according to the McDonald criteria of 2017
* First treatment during the course of MS therapy with ocrelizumab SC according to the local prescribing information, regardless of the reason for starting treatment with ocrelizumab

Exclusion Criteria:

* Participation in interventional studies investigating DMTs for MS
* Prior or simultaneous participation in CONFIDENCE or MoOzaRt (ISRCTN55332718) non interventional study (NIS) at the same study site
* Prior treatment with rituximab (MabThera®) or ublituximab (Briumvi®)
* Severe psychiatric disability
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with relapsing multiple sclerosis (RMS) and primary progressive multiple sclerosis (PPMS), diagnosed according to McDonald criteria of 2017, and treated with ocrelizumab SC for the first time during routine clinical practice will be observed in this study.
Sampling Method: Probability Sample
Enrollment: 842 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Their Level of by Satisfaction With Ocrelizumab SC After 12 Months Assessed Using TASQ-SC | Month 12
  TASQ-SC is a 12-item, participant-reported questionnaire measuring the impact of treatment administration on five domains: Physical Impact, Psychological Impact, Impact on Activities of Daily Living, Convenience, and Satisfaction. Each of the domain/scale scores is scored on a scale of 1-100, where higher scores indicate higher overall satisfaction with the therapy.

SECONDARY OUTCOMES:
Number of Participants by Their Level of Satisfaction With Ocrelizumab SC After the First Injection and After 6 Months Assessed Using TASQ-SC | Baseline, Month 6
  TASQ-SC is a 12-item, participant-reported questionnaire measuring the impact of treatment administration on five domains: Physical Impact, Psychological Impact, Impact on Activities of Daily Living, Convenience, and Satisfaction. Each of the domain/scale scores is scored on a scale of 1-100, where higher scores indicate higher overall satisfaction with the therapy.
Change From Baseline in NfL Protein Levels in Serum | Month 6, Month 12
Concentration of NfL Protein Levels in Serum | Baseline, Month 6, Month 12
Correlation Between NfL Protein Levels in Serum With MS Relapse | Up to Month 12
  The changes in levels of NfL protein levels in serum and its correlation with MS relapse will be analyzed using Pearson or Spearman correlation coefficients.
Correlation Between NfL Protein Levels in Serum With Expanded Disability Status Scale (EDSS) | Up to Month 12
  The changes in levels of NfL protein levels in serum and its correlation with EDSS will be analyzed using Pearson or Spearman correlation coefficients. EDSS is a scale for assessing neurologic impairment in MS. Values are from 0 points (normal neurological examination) up to 10 points (death), increasing in increments of 0.5 points. Higher scores represent increased disability.
Correlation Between NfL Protein Levels in Serum With Previous MS Disease Modifying Therapy (DMT) | Up to Month 12
  The changes in levels of NfL protein in serum and its correlation with DMT will be analyzed using Pearson or Spearman correlation coefficients.
Correlation Between NfL Protein Levels in Serum With NfL Confounder - Serum Creatinine | Up to Month 12
  The changes in levels of NfL protein in serum and its correlation with serum creatinine will be analyzed using Pearson or Spearman correlation coefficients.
Correlation Between NfL Protein Levels in Serum With NfL Confounder - Co-morbidities | Up to Month 12
  The changes in levels of NfL protein in serum and its correlation with co-morbidities will be analyzed using Pearson or Spearman correlation coefficients.
Correlation Between NfL Protein Levels in Serum With NfL Confounder - Age | Up to Month 12
  The changes in levels of NfL protein in serum and its correlation with age will be analyzed using Pearson or Spearman correlation coefficients.
Correlation Between NfL Protein Levels in Serum With NfL Confounder - Body Mass Index [BMI] | Up to Month 12
  The changes in levels of NfL protein in serum and its correlation with BMI will be analyzed using Pearson or Spearman correlation coefficients.
Correlation Between NfL Protein Levels in Serum With Magnetic Resonance Imaging (MRI) Lesion Count | Up to Month 12
  The changes in levels of NfL protein in serum and its correlation with MRI lesion count will be analyzed using Pearson or Spearman correlation coefficients.
Correlation Between NfL Protein Levels in Serum With Glial Fibrillary Acidic Protein (GFAP) Levels | Up to Month 12
  The changes in levels of NfL protein in serum and its correlation with GFAP levels will be analyzed using Pearson or Spearman correlation coefficients.
Correlation Between NfL Protein Levels in Serum With No Evidence of Disease Activity-3 (NEDA-3) | Up to Month 12
  NEDA-3 is defined by no confirmed MS relapse, no new or enlarging T2 lesions, no Gadolinium-positive T1 lesions, and no six-month confirmed disability worsening. The changes in levels of NfL protein in serum and its correlation with NEDA-3 will be analyzed using Pearson or Spearman correlation coefficients.
Change From Baseline in Participant Satisfaction With Ocrelizumab SC Assessed Using Treatment Satisfaction Questionnaire for Medication (TSQM) 1.4 | Month 6, Month 12
  TSQM version 1.4 is a 14-item questionnaire used to measure level of satisfaction or dissatisfaction with the medication on 4 domains: Effectiveness, Side Effects, Convenience, and Global Satisfaction. Each of the domain is scored on likert-type scales of 5 or 7 points ranging from 1 (least satisfied) to 5 or 7 (most satisfied). Item scores are summarized to give four domain scores, which are in turn transformed to a scale of 0-100. Higher scores indicate higher overall satisfaction with the therapy.
Number of Participants by Their Level of Satisfaction With Ocrelizumab SC Assessed by Physician Survey | Baseline, Month 6, Month 12
Annualized Relapse Rate | Month 12
Percentage of Participants With Progression Independent of Relapse Activity (PIRA) | Up to Month 12
Number of Participants With Non-serious Adverse Events (nsAEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interests (AESIs) | Up to Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (72):
- Germany (70):
  - Uniklinik RWTH Aachen, Aachen
  - Neuropraxis im Stadtpalais Dres. Ulzheimer/Herröder/Wessig GbR, Aschaffenburg
  - Neurologie Bad Soden, Bad Soden
  - Neurologische Praxis - Kallmann Neurologie - mszb, Bamberg
  - Neurologisches Facharztzentrum Berlin am Sankt Gertrauden-Krankenhaus, Berlin
  - NEUROZENTRUM tempelhof.berlin, Berlin
  - Praxis Dr. Said Masri, Berlin
  - Jüdisches Krankenhaus Berlin, Berlin
  - NeuroZentrum Zehlendorf Dr. Ringel und Dr. Scherer, Berlin
  - Neurologisches Zentrum für Bewegungsstörungen und Diagnostik, Berlin
  - St. Josef-Hospital, Bochum
  - Dres. Lippert/Kausch, Bogen
  - Krankenhaus Buchholz Abt. Neurologie, Buchholz
  - Neuropraxis Celle: Praxis für Neurologie & Psychatrie, Celle
  - Praxisgemeinschaft Dres. Sylke Domke und Vasil Gjaurov, Chemnitz
  - NeuroMed Campus Neurologische Gemeinschaftspraxis am St. Elisabeth Krankenhaus, Cologne
  - Gemeinschaftspraxis Dr. med. Josef Leclaire und Dr. med. Thomas Rotermund, Dortmund
  - Gemeinschaftspraxis für Neurologie, Düsseldorf
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Gemeinschaftspraxis für Neurologie und Psychiatrie, Psychotherapie, Eltville
  - NeuroCentrum Odenwald, Erbach/Odenwald
  - Universitätsklinikum Erlangen, Neurologische Klinik, Erlangen
  - Zentrum für ambulante Neurologie / Praxis Knorn Landefeld Friedrich, Essen
  - Praxis für Neurologie, Nervenheilkunde & Neurochirurgie, Forchheim
  - Universitätsklinikum Freiburg, Klinik für Neurologie und Neurophysiologie, Freiburg im Breisgau
  - Praxis im Bahnhof, Füssen
  - Neurologie & Psychiatrie Gladenbach - MS-Zentrum, Gladenbach
  - Neurologische Praxis Eppendorf, Hamburg
  - Neurologische Praxis, Hanover
  - Oberhavel Kliniken GmbH, Klinik Hennigsdorf, Neurologie, Hennigsdorf
  - Praxis Dr. Hospely, Herford
  - Haus- und Facharztzentrum Laucherttal / Alb, Hettingen
  - Klinikum Ibbenbüren gmbH, Ibbenbueren
  - Augustahospital Anholt;Neurologie, Isselburg
  - Universitätsklinikum Jena, Klinik für Neurologie, Jena
  - Arztpraxis Dr. med. Torsten Sühnel, Leipzig
  - Neurologische Praxis Dr. Ehrlich, Leipzig
  - Neurologie im Ulrichshaus Magdeburg, Magdeburg
  - Universitätsklinikum Magdeburg, Magdeburg
  - Neuroplus Dres. Lennart Thilmann/ Patrick Thilmann, Mannheim
  - Universitätsklinikum Mannheim, Mannheim
  - Universitätsklinikum Giessen und Marburg, Marburg
  - Praxis Dr. Leussink, Meerbusch
  - Neurologie am Preußenmuseum, Minden
  - Neurologie München Nord, München
  - Praxis für Neurologie und Psychiatrie am Prinzregentenplatz, München
  - Neurologisch-psychiatrische Praxis im A4, Neu-Ulm
  - Praxis Dr. med. Bergmann, Neuburg am Inn
  - Neurologie Nürnberg-Eibach, Nuremberg
  - Neurologie an der Hase, Osnabrück
  - Dres. Beckmann / Schlüter, Öhringen
  - Facharztpraxis für Neurologie und Psychiatrie Dres Mattes/Stockert, Pforzheim
  - Neurologisches Studienzentrum Artland, Quakenbrück
  - Gemeinschaftspraxis für Neurologie, Regensburg
  - Praxis Dr. Stienker-Fisse, Remscheid
  - ZNS Südpfalz, Rülzheim
  - Neurologische Praxis Dr. Wagner, Schwetzingen
  - Gemeinschaftspraxis für Neurologie, Psychiatrie und Psychotherapie, Siegen
  - Praxis für Neurologie und Psychiatrie, Siegen
  - EMSA - Zentrum für Neurologie?/?Psychiatrie?/?Neuroradiologie, Singen
  - Praxis Dr. med. Max Deist und Michael Ernst ?Sinsheim, Sinsheim
  - Gemeinschaftspraxis Dr. Wolfram von Pannwitz, MBA & Dr. med. Marie Perle Brinckmann, Steglitz
  - Praxis Dr. med. Andreas Kowalik, Arzt für Neurologie und Psychiatrie, Stuttgart
  - Sauerlandklinik Hachen, Sundern
  - Universitätsklinikum Tübingen, Zentrum für Neurologie, Tübingen
  - Nervenfachaerztliche Gemeinschaftspraxis Ulm, Ulm
  - Neuropraxis München Süd, Unterhaching
  - Praxis für Neurologie, Psychiatrie und Epileptologie, Weil der Stadt
  - Praxis Dr. Michaela Krause, Wolfratshausen
  - Heinrich-Braun-Krankenhaus Städtisches Klinikum, Zwickau
- Switzerland (2):
  - Inselspital-Universitaetsspital Bern, Bern
  - Bellevue Medical Grop AG, Zurich

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing